CLINICAL TRIAL: NCT00545454
Title: Activity and Safety of Oral Administration of SSR150106XB for the Reduction of Inflammation in Patients With Active Rheumatoid Arthritis (RA): A 4-week, Multicenter, Randomized, Double-blind, Placebo-controlled Parallel Group Study of 90 µg Administered Once Daily and 90 µg Once Every Other Day
Brief Title: Activity and Safety of Oral Administration of SSR150106XB for the Reduction of Inflammation in Patients With Active Rheumatoid Arthritis
Acronym: ACCORD-RA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACT5488; EudraCT 2007-00760-24
Record Dates: First submitted 2007-10-16; First posted 2007-10-17 (Estimated); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Rheumatoid Arthritis
Keywords: Inflammation; anti-cytokine; anti-chemokine
MeSH Terms: conditions — Arthritis, Rheumatoid; Inflammation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- SSR150106 QD (Experimental): 90 micro grams oral solution once daily (QD)
  Interventions: Drug: SSR150106
- SSR150106 OEQD (Experimental): 90 micro grams oral solution once every other day (OEQD)
  Interventions: Drug: SSR150106
- Placebo (Placebo Comparator): oral solution QD or OEQD
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: SSR150106
  Arms: SSR150106 OEQD; SSR150106 QD
Drug: Placebos
  Arms: Placebo

SUMMARY:
The primary objective of this study is to assess the reduction of systemic inflammation as measured by serum levels of C-reactive protein (CRP).

The secondary objectives are:

* to assess the reduction of systemic inflammation as measured changes in acute phase protein, serum amyloid A (SAA) and cytokine interleukin-6 (IL-6), and clinical American College of Rheumatology response rate, and morning stiffness duration;
* to assess the effect on pain relief within first 14 days;
* to obtain evidence of the safety and tolerability of SSR150106;
* to document trough plasma levels of SSR150106 and its first metabolite.

ELIGIBILITY:
Inclusion Criteria:

* Either treatment-naïve patients, or those who have discontinued their Rheumatoid Arthritis-directed medication due to intolerability or insufficient efficacy
* At least 9 out of 68 tender joints; 6 out of 66 swollen joints; morning stiffness 45 min
* C-Reactive Protein >=1.8 mg/dl confirmed during screening period
* Non-poor Cytochrome P2D6 metabolizer status

Exclusion Criteria:

* Functional Rheumatoid Arthritis class IV
* Fever
* Infections with hepatitis B, or C, or HIV
* Presence or history (<5 years) of cancer
* Manifest or latent tuberculosis
* Functional abnormalities (including laboratory values) judged as clinically relevant

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2007-10; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in mean C-Reactive Protein level | end of the 4-week double-blind treatment period

SECONDARY OUTCOMES:
C-Reactive Protein, Serum Amyloid A and Cytokine Interleukin-6 levels | at all time points measured
Improvement responder rates based on the American College of Rheumatology criteria | at all time points measured
Pain relief (change from baseline) | until day 14
Safety and tolerability | During the entire study patient's participation
Plasma levels of SSR150106 and its first metabolite | On a weekly basis during treatment phase, except at the end of the 3rd week

CONTACTS AND LOCATIONS:
Overall Officials: Karel PAVELKA, Prof., MD, Principal Investigator — Karel PAVELKA
Locations (7):
- Sanofi-Aventis Administrative Office, Sofia, Bulgaria
- Sanofi-Aventis Administrative Office, Zagreb, Croatia
- Sanofi-Aventis Administrative Office, Prague, Czechia
- Sanofi-Aventis Administrative Office, Bucharest, Romania
- Sanofi-Aventis Administrative Office, Moscow, Russia
- Sanofi-Aventis Administrative Office, Bratislava, Slovakia
- Sanofi-Aventis Administrative Office, Kiev, Ukraine

REFERENCES:
- See also: Related Info — http://www.sanofi-aventis.com